CLINICAL TRIAL: NCT03200366
Title: Comparing Interventions to Increase Colorectal Cancer Screening in Low-Income and Minority Patients
Brief Title: Comparing Interventions to Increase Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Susan Rawl, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1605880142; IHS-1507-31333 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
Keywords: Cancer Screening Tests; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored DVD (Active Comparator): Tailored digital video disc (DVD)
  Interventions: Behavioral: Tailored DVD
- Tailored DVD + Patient Navigation (Active Comparator): Tailored digital video disc (DVD) plus Patient Navigation by a population health nurse in the healthcare system
  Interventions: Behavioral: Tailored DVD; Behavioral: Patient Navigation
- Usual Care (No Intervention): Care normally provided by a nurse in the endoscopy department of the healthcare system

INTERVENTIONS:
Behavioral: Tailored DVD — A 20 minute tailored DVD titled "Approaches to Colon Testing" is viewed by participants. It is designed to encourage CRC screening uptake by colonoscopy or FIT by increasing the participant's CRC knowledge and beliefs about the benefits of screening, reducing barriers to screening, and increasing self-efficacy for screening by demonstrating how these tests are performed.
  Arms: Tailored DVD; Tailored DVD + Patient Navigation
Behavioral: Patient Navigation — Participants talk by telephone with a Patient Navigator who is a trained nurse. The Patient Navigator determines if participants viewed the tailored DVD and answers any questions about the content. The Patient Navigator then provides telephone counseling on CRC and screening tests to: (1) increase knowledge, perceived benefits, and self-efficacy; (2) reduce barriers; (3) enhance access; and (4) provide social support.
  Arms: Tailored DVD + Patient Navigation

SUMMARY:
The purpose of this study is to test different approaches to help people understand the purpose of colorectal cancer (CRC) screening, two screening test options available, and the barriers to screening so they can make informed decisions about CRC screening. Participants will be randomly assigned to one of three groups: (1) one group will receive a tailored digital video disc (DVD) in the mail; (2) another group will receive the mailed DVD plus telephone calls from a patient navigator; and (3) the third group will receive the care normally provided by the healthcare system's endoscopy department.

The investigators hypothesize the following: (1) participants who receive the tailored DVD plus the patient navigation intervention will have higher rates of CRC screening with the fecal immunochemical test (FIT), colonoscopy, or either screening test compared to those who receive the tailored DVD alone; (2) participants who receive either intervention (DVD only or DVD plus patient navigation) will have higher rates of CRC screening with FIT, colonoscopy, or either screening test than those who receive usual care; and (3) participants who receive either intervention who complete colonoscopy will have better quality of bowel preparation, less anxiety about the procedure, and greater satisfaction with the colonoscopy experience than those who receive usual care.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) often can be prevented through regular screening and although multiple screening tests are available, colonoscopy is often the only screening test offered to patients. Unfortunately, up to half of people in some hospitals who receive a recommendation and are scheduled for colonoscopy do not complete the test. Reasons for not completing colonoscopy include lack of awareness of the need for, and benefits of, screening, fear of pain, fear of finding cancer, unpleasantness of the bowel preparation, cost, transportation issues, and the unwillingness to undergo an invasive test in the absence of symptoms. The process of bowel cleansing is one of the most challenging aspects of having a colonoscopy. Interventions that improve patients' knowledge about CRC screening, including test options other than colonoscopy, enhance access, improve skills needed to complete CRC screening, and reduce barriers will lead to greater numbers of people being screened. Patient navigation and computer tailored interventions have been shown to be effective approaches to increase CRC and other cancer screening but there is no evidence of their comparative effectiveness. The purpose of this study is to compare two health system-based interventions, with one another and with usual care, to increase completion rates among a diverse sample of patients. The investigators will enroll an ethnically diverse group of 450 men and women aged 50-75,or aged 45-75 if African American, who are at average risk for CRC and were referred and scheduled for colonoscopy at one endoscopy department but canceled or did not attend their scheduled appointment. Participants will be randomized to receive: (1) a mailed tailored digital video disc (DVD) alone; 2) the mailed tailored DVD plus a telephone-based Patient Navigator; or 3) usual care. Data will be collected at baseline, at 6 months and at 9 months post-baseline. Interviews to assess receipt, viewing, and satisfaction with the tailored DVD will be conducted 2 weeks after mailing. Satisfaction with the patient navigator will be assessed at 6 months. Multivariable logistic regression analyses will be used to test the interventions' effects on CRC screening test completion and, for those who complete colonoscopy, quality of bowel preparation. The investigators will also examine whether these interventions change knowledge about CRC and screening as well as health beliefs (perceived risk, perceived benefits, barriers, and self-efficacy) about screening. From this study, the investigators will learn how effective these two standardized, easy to disseminate health system-based interventions are compared to each other and to usual care. If the interventions are found to be equally effective, or differentially effective for different subgroups of patients, healthcare systems may consider implementing one or both of these interventions in their settings.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a screening colonoscopy that was not done (i.e, canceled or no show)

Exclusion Criteria:

* Unable to speak, read, and write English
* Personal history of CRC or polyps
* Personal history of conditions that place participants at high risk for CRC such as ulcerative colitis, Crohn's disease, or known hereditary syndromes such as familial adenomatous polyposis or hereditary nonpolyposis colorectal cancer
* Family history of CRC which increases the participant's risk for CRC
* Advised by a health care provider to not have a colonoscopy due to the participant's health
* Speech impairment
* Hearing impairment
* Cognitive impairment
* Vision impairment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Rawl, PhD,RN, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University School of Nursing, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
A copy of the complete, cleaned, de-identified data set used to conduct the final analyses will be made available in SAS and SPSS formats.
Supporting Information: Study Protocol, SAP
Time Frame: Available by September 30, 2021
Access Criteria: Request in writing to the the study's Principal Investigator, Dr. Susan Rawl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 371 primary care patients from Eskenazi Health clinics located ln Indianapolis, Indiana. Participants were recruited between July 2017 to November 2019. Participants were enrolled after providing informed consent and HIPAA authorization to obtain CRC screening information from their electronic medical record (EMR). EMR was reviewed for completion of CRC screening by colonoscopy and FIT for ALL participants, regardless of whether or not post-baseline interviews were completed.
Groups:
- Tailored DVD: Tailored digital video disc (DVD)
  DVD: A 20 minute tailored DVD titled "Approaches to Colon Testing" is viewed by participants. It is designed to encourage CRC screening uptake by colonoscopy or FIT by increasing the participant's CRC knowledge and beliefs about the benefits of screening, reducing barriers to screening, and increasing self-efficacy for screening by demonstrating how these tests are performed.
- Tailored DVD + Patient Navigation: Tailored digital video disc (DVD) plus Patient Navigation by a population health nurse in the healthcare system
  DVD: A 20 minute tailored DVD titled "Approaches to Colon Testing" is viewed by participants. It is designed to encourage CRC screening uptake by colonoscopy or FIT by increasing the participant's CRC knowledge and beliefs about the benefits of screening, reducing barriers to screening, and increasing self-efficacy for screening by demonstrating how these tests are performed.
  Patient Navigation: Participants talk by telephone with a Patient Navigator who is a trained nurse. The Patient Navigator determines if participants viewed the tailored DVD and answers any questions about the content. The Patient Navigator then provides telephone counseling on CRC and screening tests to: (1) increase knowledge, perceived benefits, and self-efficacy; (2) reduce barriers; (3) enhance access; and (4) provide social support.
Period: Baseline Interview With Randomization
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Started | 123 | 120 | 128
Completed | 123 | 120 | 128
Not Completed | 0 | 0 | 0
Period: Tailored DVD Intervention Given
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Started | 123 | 120 | 0
Completed (Tailored DVD mailed 1-2 days post-randomization to participants in the 2 intervention arms: Tailored DVD and Tailored DVD + Patient Navigation. DVD was NOT mailed to participants in Usual Care arm.) | 123 | 120 | 0
Not Completed | 0 | 0 | 0
Period: Patient Navigation Intervention Given
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Started (Patient Navigation delivered from 2 weeks post-randomization up to 6 months post-randomization to only participants in Tailored DVD + Patient Navigation arm.) | 0 | 120 | 0
Completed | 0 | 89 | 0
Not Completed | 0 | 31 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 25 | 0
Not completed — Not attempted/missed by nurse | 0 | 1 | 0
Not completed — Colonoscopy already re-scheduled and completed | 0 | 2 | 0
Not completed — Declined navigation intervention | 0 | 1 | 0
Period: 6 Month Post-Baseline Interview
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Started ("Started" number excludes 2 participants in Tailored DVD +Patient Navigation arm that were deceased before 6 month post-baseline timepoint.) | 123 | 118 | 128
Completed | 93 | 95 | 109
Not Completed | 30 | 23 | 19
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 27 | 21 | 17
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Refused 6 month interview but continued in study | 1 | 0 | 0
Not completed — Not attempted/missed by data collectors | 0 | 0 | 1
Period: 9 Month Post-Baseline Interview
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Started ("Started" number excludes participants that were deceased or withdrawn before 9 month post-baseline timepoint: Tailored DVD arm n=2; Tailored DVD + Patient Navigation arm n=4; and Usual Care arm n=1.) | 121 | 116 | 127
Completed | 97 | 95 | 116
Not Completed | 24 | 21 | 11
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 23 | 18 | 9
Not completed — Withdrawal by PI | 0 | 0 | 1
Not completed — Refused interview | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care | Total
Number analyzed (Participants) | 123 | 120 | 128 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (6.07) | 57.29 (5.63) | 57.83 (6.17) | 57.78 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 73 | 77 | 225
  Male | 48 | 47 | 51 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Whte | 35 | 33 | 36 | 104
  Non-Hispanic Non-White | 83 | 82 | 87 | 252
  Other | 5 | 5 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 123 | 120 | 128 | 371
Married/Partnered [Count of Participants; unit: Participants] — Participants who are either married or living with a partner. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant from the Tailored DVD + Patient Navigation group whose data were missing.
  Participants
    number analyzed (Participants) | 123 | 119 | 128 | 370
    (all) | 38 | 36 | 40 | 114
Education [Count of Participants; unit: Participants] — Participants highest grade or year of school completed. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 123 | 120 | 127 | 370
    No school through 11th grade | 28 | 22 | 35 | 85
    12th grade, high school, diploma, or GED | 42 | 41 | 46 | 129
    Vocational school or 1-3 years college | 39 | 45 | 34 | 118
    4 year college graduate, some graduate work, or completed graduate degree | 14 | 12 | 12 | 38
Number in Household [Count of Participants; unit: Participants] — Number of persons, including the participant, who live in their household. Population: Enrolled participants who completed the baseline interview. Excludes 2 participants in the Tailored DVD group whose data were missing. Excludes 3 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 2 participants in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 121 | 117 | 126 | 364
    1 person | 47 | 39 | 52 | 138
    2 persons | 46 | 44 | 33 | 123
    3 or more persons | 28 | 34 | 41 | 103
Children Under Age 18 in Household [Count of Participants; unit: Participants] — Participants with children younger than 18 living in their household. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 1 participant in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 123 | 119 | 127 | 369
    (all) | 20 | 25 | 33 | 78
Employment Status [Count of Participants; unit: Participants] — Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 123 | 120 | 127 | 370
    Not employed | 83 | 66 | 87 | 236
    Part-time | 18 | 19 | 16 | 53
    Full-time | 22 | 35 | 24 | 81
Household Income [Count of Participants; unit: Participants] — Total combined yearly household income before taxes. Population: Enrolled participants who completed the baseline interview. Excludes 2 participants in the Tailored DVD group whose data were missing. Excludes 6 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 5 participants in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 121 | 114 | 123 | 358
    Less than $15,000 | 57 | 45 | 52 | 154
    $15,001-$30,000 | 46 | 40 | 44 | 130
    $30,001-$50,000 | 13 | 20 | 15 | 48
    $50,001 to more than $100,000 | 5 | 9 | 12 | 26
Household Income Categorized by $15K Level [Count of Participants; unit: Participants] — Total combined yearly household income before taxes, categorized as below $15,000 vs. $15,000 or more. Population: Enrolled participants who completed the baseline interview. Excludes 2 participants in the Tailored DVD group whose data were missing. Excludes 6 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 5 participants in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 121 | 114 | 123 | 358
    Less than $15,000 | 57 | 45 | 52 | 154
    $15,000 or more | 64 | 69 | 71 | 204
Adequacy of Income [Count of Participants; unit: Participants] — Participants described the adequacy of their household income to pay for things. Population: Enrolled participants who completed the baseline interview. Excludes 4 participants in the Tailored DVD group whose data were missing. Excludes 7 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 6 participants in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 119 | 113 | 122 | 354
    After paying the bills, there is enough money for special things that the participant wants. | 17 | 16 | 20 | 53
    There is enough money to pay the bills, but little spare money to buy extra or special things. | 44 | 41 | 44 | 129
    There is enough money to pay the bills, but only because the participant cuts back on things. | 22 | 22 | 21 | 65
    The participant has difficulty paying the bills, no matter what is done. | 36 | 34 | 37 | 107
Health Insurance Coverage [Count of Participants; unit: Participants] — Participants covered by health insurance or some other kind of health care plan. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in the Usual Care group whose data were missing.
  Participants
    number analyzed (Participants) | 123 | 120 | 127 | 370
    (all) | 114 | 114 | 121 | 349
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is an estimate of body fat that is calculated using participants self report of height and weight. BMI values are correlated with weight categories. A BMI <18.5 means underweight; BMI=18.5-24.9 means normal weight; BMI=25.0-29.9 means overweight; and BMI > 30 means obese. A high BMI is associated with an increased risk for chronic diseases such as heart disease, high blood pressure, and type 2 diabetes. Population: Enrolled participants who completed the baseline interview. Excludes 3 participants in the Tailored DVD + Patient Navigation group whose data were missing.
  kg/m^2
    number analyzed (Participants) | 123 | 117 | 128 | 368
    (all) | 31.57 (8.89) | 30.18 (7.86) | 31.50 (8.93) | 31.10 (8.59)
Global Physical Health [Mean (Standard Deviation); unit: units on a scale] — Global physical health status was measured using the subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS) validated instrument. The subscale uses 4 items and measures general physical health, physical functioning, pain, and fatigue. Response options range from 1=poor to 5=excellent. Scores range from a minimum of 4 to a maximum of 20. Higher scores indicate better physical health. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 3 participants in the Usual Care group whose data were missing.
  units on a scale
    number analyzed (Participants) | 123 | 119 | 125 | 367
    (all) | 12.64 (3.24) | 13.37 (3.29) | 12.89 (3.38) | 12.96 (3.31)
Global Mental Health [Mean (Standard Deviation); unit: units on a scale] — Global mental health status was measured using the subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS) validated instrument. The subscale uses 4 items and measures quality of life, general mental health, satisfaction with social activities/relationships, and emotional problems. Response options range from 1=poor to 5=excellent. Scores range from a minimum of 4 to a maximum of 20. Higher scores indicate better mental health. Population: Enrolled participants who completed the baseline interview. Excludes 2 participants in the Tailored DVD + Patient Navigation group whose data were missing.
  units on a scale
    number analyzed (Participants) | 123 | 118 | 128 | 369
    (all) | 12.86 (3.19) | 12.73 (3.50) | 12.88 (3.31) | 12.82 (3.32)
Health Literacy [Mean (Standard Deviation); unit: units on a scale] — Health literacy was measured using Chew's Brief Health Literacy Screen validated instrument. This 3-item scale assesses participants' confidence in filling out medical forms independently, if they need help from others to read hospital materials, and if they have problems learning about their medical condition because of difficulty understanding written information. Recoded response options range from 1=no confidence/always need help/always difficult to 5=extremely confident/never need help/never difficult. Scores range from 3 to 15. Higher scores indicate greater health literacy. Population: Enrolled participants who completed the baseline interview. Excludes 1 participant in the Tailored DVD + Patient Navigation group whose data were missing.
  units on a scale
    number analyzed (Participants) | 123 | 119 | 128 | 370
    (all) | 12.20 (2.74) | 11.97 (2.64) | 11.91 (3.18) | 12.03 (2.87)
Comorbidity [Mean (Standard Deviation); unit: units on a scale] — Comorbidity was measured by self-report using Sangha's comordibity questionnaire. Twelve common health problems (heart disease, high blood pressure, diabetes, etc.) are assessed by asking participants if they ever had the problem, if they currently receive treatment for it, and if it currently limits their activities. Each question is scored as yes=1 or no=0 resulting in a possible score of 0 to 3 per health problem. Scale scores range from 0 to 36. Higher scale scores indicate greater comorbidity.
  units on a scale | 8.24 (4.86) | 7.73 (4.83) | 7.56 (4.72) | 7.84 (4.80)
Knowledge of CRC and Screening [Mean (Standard Deviation); unit: units on a scale] — Knowledge of CRC and screening is measured by self-report using a 9-item multidimensional scale. Each item is scored as 1=correct or 0=incorrect, summed to yield a scale score, and the mean calculated. Scores range from 0 to 9. Higher scale scores and means indicate greater knowledge of CRC and screening tests.
  units on a scale | 3.54 (1.83) | 3.62 (1.77) | 2.93 (1.72) | 3.36 (1.80)
Perceived Risk for CRC [Mean (Standard Deviation); unit: units on a scale] — Perceived risk for CRC is measured by self-report using a 3-item scale. We ask participants how likely it is that they will get colon cancer sometime during their lifetime, within the next 10 years, and within the next 5 years. Each item is scored from 1 to 4 (1=very unlikely; 4=very likely) and the mean of the 3 items calculated. Higher mean scores indicate a greater perceived risk for getting CRC. Population: Enrolled participants who completed the baseline interview. Excludes 9 participants in the Tailored DVD group whose data were missing. Excludes 2 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 4 participants in the Usual Care group whose data were missing.
  units on a scale
    number analyzed (Participants) | 114 | 118 | 124 | 356
    (all) | 1.97 (0.73) | 1.94 (0.80) | 2.03 (0.81) | 1.98 (0.78)
Colonoscopy Stage of Adoption [Count of Participants; unit: Participants] — Participants staged in terms of their readiness screen for CRC by having a colonoscopy. If not planning to have a colonoscopy in the next 6 months, staging was precontemplation. If planning to have a colonoscopy in the next 6 months, but no appointment scheduled, staging was contemplation. If an appointment was scheduled to have a colonoscopy within the next 6 months, staging was preparation.
  Participants
    Precontemplation | 27 | 25 | 29 | 81
    Contemplation | 70 | 67 | 61 | 198
    Preparation | 26 | 28 | 38 | 92
Colonoscopy-Related Procedural Anxiety [Mean (Standard Deviation); unit: units on a scale] — Colonoscopy-related procedural anxiety is measured by self-report using the 6-item short form of the State Anxiety Scale of the State-Trait Anxiety Inventory. Each item is scored from 1 to 4 (1=not at all; 4=very much so) and the mean of the 4 items calculated. Higher mean scores indicate greater anxiety. Population: Excludes 1 participant in the Tailored DVD group whose data were missing.
  units on a scale
    number analyzed (Participants) | 122 | 120 | 128 | 370
    (all) | 2.59 (0.68) | 2.60 (0.69) | 2.52 (0.59) | 2.57 (0.65)
Perceived Benefits of CRC Screening by Colonoscopy [Mean (Standard Deviation); unit: units on a scale] — Perceived benefits of CRC screening by colonoscopy is measured by self-report using a 4-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 4 items calculated. Higher mean scores indicate greater perceived benefits of screening by colonoscopy. Population: Enrolled participants who completed the baseline interview. Excludes 2 participants in the Tailored DVD group whose data was missing. Excludes 1 participant in the Tailored DVD + Patient Navigation group whose data was missing.
  units on a scale
    number analyzed (Participants) | 121 | 119 | 128 | 368
    (all) | 3.22 (0.61) | 3.31 (0.57) | 3.27 (0.56) | 3.27 (0.58)
Perceived Barriers to CRC Screening by Colonoscopy [Mean (Standard Deviation); unit: units on a scale] — Perceived barriers to colonoscopy is measured by self-report using a 16-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 16 items calculated. Higher mean scores indicate greater perceived barriers to screening by colonoscopy.
  units on a scale | 2.21 (0.56) | 2.33 (0.55) | 2.29 (0.62) | 2.28 (0.58)
Perceived Self-Efficacy for CRC Screening by Colonoscopy [Mean (Standard Deviation); unit: units on a scale] — Perceived self-efficacy for colonoscopy is measured by self-report using an 11-item scale. Each item is scored from 1 to 4 (1=not at all sure; 4=very sure) and the mean of the 11 items calculated. Higher mean scores indicate greater perceived self-efficacy for CRC screening by colonoscopy.
  units on a scale | 3.33 (0.56) | 3.33 (0.49) | 3.36 (0.55) | 3.34 (0.53)
Fecal Immunochemical Test Stage of Adoption [Count of Participants; unit: Participants] — Participants staged in terms of their readiness to adopt an at-home fecal immunochemical test (FIT) to screen for CRC. If not planning to do a FIT in the next 6 months, staging was precontemplation. If planning to do a FIT in the next 6 months, but did not have a FIT kit at home, staging was contemplation. If planning to do a FIT within the next 6 months and had a FIT kit at home, staging was preparation. If a FIT was already done within the last 12 months, staging was action.
  Participants
    Precontemplation | 73 | 80 | 87 | 240
    Contemplation | 23 | 20 | 20 | 63
    Preparation | 3 | 8 | 6 | 17
    Action | 24 | 12 | 15 | 51
Perceived Benefits of CRC Screening by FIT [Mean (Standard Deviation); unit: units on a scale] — Perceived benefits of CRC screening by FIT is measured by self-report using a 3-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 3 items calculated. Higher mean scores indicate greater perceived benefits of screening by FIT. Population: Enrolled participants who completed the baseline interview. Excludes 6 participants in the Tailored DVD group whose data were missing. Excludes 3 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 2 participants in the Usual Care group whose data were missing.
  units on a scale
    number analyzed (Participants) | 117 | 117 | 126 | 360
    (all) | 3.06 (0.73) | 3.15 (0.64) | 3.16 (0.70) | 3.13 (0.69)
Perceived Barriers to CRC Screening by FIT [Mean (Standard Deviation); unit: units on a scale] — Perceived barriers to FIT is measured by self-report using a 10-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 10 items calculated. Higher mean scores indicate greater perceived barriers to screening by FIT.
  units on a scale | 1.97 (0.55) | 2.20 (0.57) | 2.11 (0.62) | 2.10 (0.59)
Perceived Self-Efficacy for CRC Screening by FIT [Mean (Standard Deviation); unit: units on a scale] — Perceived self-efficacy for FIT is measured by self-report using a 7-item scale. Each item is scored from 1 to 4 (1=not at all sure; 4=very sure) and the mean of the 7 items calculated. Higher mean scores indicate greater perceived self-efficacy for CRC screening by FIT.
  units on a scale | 3.63 (0.49) | 3.59 (0.48) | 3.63 (0.47) | 3.61 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Participants Completing CRC Screening Per Electronic Medical Record Documentation
Description: Number of participants completing CRC screening by any test (defined as colonoscopy or FIT) is measured by electronic medical record review. Dates that participants had a colonoscopy and dates of FIT analysis are extracted from the electronic medical record.
Time Frame: 12 months post-baseline interview
Population: All enrolled participants who completed the baseline interview and were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 123 | 120 | 128
Participants | 37 | 59 | 27

2. Secondary Outcome: Participants Completing Colonoscopy Per Electronic Medical Record Documentation
Description: Number of participants completing a colonoscopy is measured by electronic medical record review (EMR). Dates that participants completed a colonoscopy are extracted from the EMR.
Time Frame: 12 months post-baseline interview
Population: All enrolled participants who completed the baseline interview and were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 123 | 120 | 128
Participants | 24 | 46 | 20

3. Secondary Outcome: Bowel Preparation Quality Rating Using Boston Bowel Preparation Scale
Description: Participants quality of bowel preparation is measured by the endoscopist during their colonoscopy procedure using the Boston Bowel Preparation Scale (BBPS). BBPS scores the total quality on a 10 point scale from 0-9. Higher scores indicate better quality of bowel preparation.
Time Frame: 12 months post-baseline interview
Population: All participants who completed a colonoscopy per EMR documentation. Analysis excludes 1 participant in Usual Care group whose BBPS score was missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 24 | 46 | 19
score on a scale | 7.13 (1.90) | 6.59 (2.40) | 7.05 (2.44)

4. Secondary Outcome: Participants With Adequate Quality of Bowel Preparation Per Modified Aronchick Rating Scale
Description: Participants quality of bowel preparation is measured by the endoscopist during their colonoscopy using a modification of the Aronchick rating scale. The Aronchick scale rates quality as 1=excellent, 2=good, 3=fair, or 4=poor. Some endoscopists choose to grade quality more generally as adequate vs. inadequate. To accommodate this variation, bowel preparation ratings have been dichotomized into adequate (excellent, good, fair, or adequate ratings) vs. inadequate (poor or inadequate ratings). Adequate is scored as 1 and indicates better quality of bowel preparation than inadequate which is scored as 0.
Time Frame: 12 months post-baseline interview
Population: All participants who completed a colonoscopy per EMR documentation.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 24 | 46 | 20
Participants | 22 | 39 | 18

5. Secondary Outcome: Colonoscopy-Related Procedural Anxiety for Participants Completing a Colonoscopy
Description: Colonoscopy-related procedural anxiety is measured by self-report using the 6-item short form of the State Anxiety Scale of the State-Trait Anxiety Inventory. Each item is scored from 1 to 4 (1=not at all; 4=very much so) with higher scores indicating greater anxiety.
Time Frame: 12 months post-baseline interview
Population: Participants who completed a colonoscopy within 12 months of the baseline interview per EMR documentation and self-reported on colonoscopy-related anxiety during the 6 or 9 month post-baseline interview. Excludes 6 participants in the Tailored DVD group whose anxiety data were missing. Excludes 6 participants in the Tailored DVD + Patient Navigation group whose anxiety data were missing. Excludes 4 participants in the Usual Care group whose anxiety data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 16 | 40 | 15
units on a scale | 2.46 (0.78) | 2.23 (0.67) | 2.28 (0.76)

6. Secondary Outcome: Satisfaction With Colonoscopy Experience
Description: Satisfaction with the colonoscopy experience is measured by self-report using a single item developed by the research team. Satisfaction is rated from 1 to 4 where 1=not at all satisfied, 2=a little satisfied, 3=mostly satisfied, and 4=completely satisfied. Scores range from 1 to 4 with higher scores indicating greater satisfaction.
Time Frame: 12 months post-baseline interview
Population: Participants who completed a colonoscopy within 12 months of the baseline interview per EMR documentation and self-reported their satisfaction with the experience during the 6 or 9 month post-baseline interview. Excludes 6 participants in the Tailored DVD group whose satisfaction data were missing. Excludes 6 participants in the Tailored DVD + Patient Navigation group whose satisfaction data were missing. Excludes 4 participants in the Usual Care group whose satisfaction data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 16 | 40 | 15
units on a scale | 3.38 (0.96) | 3.60 (0.78) | 3.13 (1.06)

7. Secondary Outcome: Participants Completing a Fecal Immunochemical Test (FIT) Per Electronic Medical Record Documentation
Description: Number of participants completing a FIT is measured by electronic medical record review (EMR). Dates of FIT analysis are extracted from the EMR.
Time Frame: 12 months post-baseline interview
Population: All enrolled participants who completed the baseline interview and were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 123 | 120 | 128
Participants | 15 | 13 | 8

8. Secondary Outcome: Participants Who Self-Reported Completing CRC Screening
Description: Number of participants who reported completing CRC screening by any test (defined as colonoscopy or FIT) during the 6 or 9 month post-baseline telephone interview.
Time Frame: 6-9 months post-baseline interview
Population: CRC screening self-reported during the 6 or 9 month follow-up telephone interview. Excludes 1 participant in Tailored DVD group due to data being collected outside of interview window. Excludes 1 participant in Usual Care group due to data being contradictory/invalid.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 101 | 103 | 117
Participants | 48 | 59 | 43

9. Secondary Outcome: Participants Who Self-Reported Completing a Colonoscopy
Description: Number of participants who reported completing a colonoscopy during the 6 or 9 month post-baseline telephone interview.
Time Frame: 6-9 months post-baseline interview
Population: Colonoscopy completed per self-report during the 6 or 9 month follow-up telephone interview. Excludes 1 participant in Tailored DVD group due to data being collected outside of interview window. Excludes 1 participant in Usual Care group due to data being contradictory/invalid.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 101 | 103 | 117
Participants | 26 | 46 | 27

10. Secondary Outcome: Participants Who Self-Reported Completing a Fecal Immunochemical Test (FIT)
Description: Number of participants who reported completing a FIT during the 6 or 9 month post-baseline telephone interview.
Time Frame: 6-9 months post-baseline interview
Population: FIT completed per self-report during the 6 or 9 month follow-up telephone interview. Excludes 1 participant in Tailored DVD group due to data being collected outside of interview window. Excludes 1 participant in Usual Care group due to data being contradictory/invalid.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 101 | 103 | 117
Participants | 34 | 28 | 20

11. Secondary Outcome: Change in Knowledge of CRC and Screening
Description: Change from baseline in knowledge of CRC and screening is measured at 6 months by self-report using a 9-item multidimensional scale. Each item is scored as 1=correct or 0=incorrect and summed to yield a scale score. Scores range from 0 to 9 with higher summated scores indicating greater knowledge of CRC and screening tests. The mean of the 9 items is calculated at baseline and 6 months post-baseline. Change from baseline equals the mean at 6 months minus the mean at baseline. Change can range from -9 to 9 with positive values indicating an increase in knowledge.
Time Frame: 6 months post-baseline interview
Population: Enrolled participants who completed the 6 month post-baseline interview. Excludes 1 participant in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 1 participant in the Usual Care group due to the data being contradictory/invalid.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 93 | 94 | 108
score on a scale | 1.14 (0.24) | 1.32 (0.25) | 0.75 (0.23)

12. Secondary Outcome: Change in Perceived Risk for CRC
Description: Change from baseline in perceived risk for CRC is measured by self-report at 6 months using a 3-item scale. We ask participants how likely it is that they will get colon cancer sometime during their lifetime, within the next 10 years, and within the next 5 years. Each item is scored from 1 to 4 (1=very unlikely; 4=very likely). Higher scores indicate a higher perceived risk for getting CRC. The mean of the 3 items is calculated at baseline and 6 months. Change in perceived risk equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in perceived risk for getting CRC.
Time Frame: 6 months post-baseline interview
Population: Enrolled participants who completed the 6 month post-baseline interview. Excludes 7 participants in the Tailored DVD group whose data were missing. Excludes 5 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 8 participants in the Usual Care group whose data were missing and 1 participant in the Usual Care group due to the data being contradictory/invalid.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 86 | 90 | 100
units on a scale | 0.23 (0.11) | 0.03 (0.11) | 0.18 (0.11)

13. Secondary Outcome: Change in Colonoscopy-Related Procedural Anxiety Regardless of Whether or Not Participants Had a Colonoscopy
Description: Change from baseline in colonoscopy-related procedural anxiety is measured at 6 months by self-report using the 6-item short form of the State Anxiety Scale of the State-Trait Anxiety Inventory. Each item is scored from 1 to 4 (1=not at all; 4=very much so) with higher scores indicating greater anxiety. The mean of the 6 items is calculated at baseline and 6 months post-baseline. Change from baseline is the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in anxiety.
Time Frame: 6 months post-baseline interview
Population: Participants who self-reported their colonoscopy-related anxiety during the 6 month post-baseline interview, regardless of their colonoscopy completion status. Excludes 1 participant in the Tailored DVD group whose data was missing. Excludes 2 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 2 participants in the Usual Care group due to data being missing for 1 participant and data being contradictory/invalid for 1 participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 92 | 93 | 107
units on a scale | -0.13 (0.09) | -0.23 (0.10) | -0.05 (0.09)

14. Secondary Outcome: Change in Perceived Benefits of CRC Screening by Colonoscopy
Description: Change from baseline in perceived benefits of CRC screening by colonoscopy is measured at 6 months by self-report using a 4-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 4 items calculated. Higher mean scores indicate greater perceived benefits of screening by colonoscopy. Change in perceived benefits equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in perceived benefits of screening by colonoscopy.
Time Frame: 6 months post-baseline interview
Population: Enrolled participants who completed the 6 month post-baseline interview. Excludes 3 participants in the Tailored DVD group whose data was missing. Excludes 2 participants in the Tailored DVD + Patient Navigation group whose data was missing. Excludes 2 participants in the Usual Care group due to data being missing for 1 participant and data being contradictory/invalid for 1 participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 90 | 93 | 107
units on a scale | 0.18 (0.08) | 0.16 (0.08) | 0.04 (0.08)

15. Secondary Outcome: Change in Perceived Barriers to CRC Screening by Colonoscopy
Description: Change from baseline in perceived barriers to CRC screening by colonoscopy is measured at 6 months by self-report using a 16-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 16 items calculated. Higher mean scores indicate greater perceived barriers to screening by colonoscopy. Change in perceived barriers equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with negative values indicating a decrease in perceived barriers to screening by colonoscopy.
Time Frame: 6 months post-baseline interview
Population: Enrolled participants who completed the 6 month post-baseline interview. Excludes 1 participant in the Tailored DVD group whose data were missing. Excludes 2 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 1 participant in Usual Care group due to data being contradictory/invalid.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 92 | 93 | 108
units on a scale | -0.21 (0.08) | 0.01 (0.09) | -0.15 (0.08)

16. Secondary Outcome: Change in Perceived Self-Efficacy for CRC Screening by Colonoscopy
Description: Change from baseline in perceived self-efficacy for colonoscopy is measured at 6 months by self-report using an 11-item scale. Each item is scored from 1 to 4 (1=not at all sure; 4=very sure) and the mean of the 11 items calculated. Higher mean scores indicate greater perceived self-efficacy for screening by colonoscopy. Change in perceived self-efficacy equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in perceived self-efficacy for screening by colonoscopy.
Time Frame: 6 months post-baseline interview
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 92 | 93 | 108
units on a scale | 0.15 (0.07) | 0.20 (0.08) | 0.06 (0.07)

17. Secondary Outcome: Change in Perceived Benefits of CRC Screening by FIT
Description: Change from baseline in perceived benefits of CRC screening by FIT is measured at 6 months by self-report using a 3-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 3 items calculated. Higher mean scores indicate greater perceived benefits of screening by FIT. Change in perceived benefits equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in perceived benefits for screening by FIT.
Time Frame: 6 months post-baseline interview
Population: Enrolled participants who completed the 6 month post-baseline interview. Excludes 6 participants in the Tailored DVD group whose data were missing. Excludes 5 participants in the Tailored DVD + Patient Navigation group whose data were missing. Excludes 2 participants in the Usual Care group whose data were missing and 1 participant in Usual Care group due to data being contradictory/invalid.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 87 | 90 | 106
units on a scale | 0.08 (0.10) | 0.07 (0.11) | -0.02 (0.10)

18. Secondary Outcome: Change in Perceived Barriers to CRC Screening by FIT
Description: Change from baseline in perceived barriers to CRC screening by FIT is measured at 6 months by self-report using a 10-item scale. Each item is scored from 1 to 4 (1=strongly disagree; 4=strongly agree) and the mean of the 10 items calculated. Higher mean scores indicate greater perceived barriers to screening by FIT. Change in perceived barriers equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with negative values indicating a decrease in perceived barriers to screening by FIT.
Time Frame: 6 months post-baseline interview
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 92 | 93 | 108
units on a scale | -0.18 (0.09) | -0.11 (0.09) | -0.16 (0.09)

19. Secondary Outcome: Change in Perceived Self-Efficacy for CRC Screening by FIT
Description: Change from baseline in perceived self-efficacy for CRC screening by FIT is measured at 6 months by self-report using a 7-item scale. Each item is scored from 1 to 4 (1=not at all sure; 4=very sure) and the mean of the 7 items calculated. Higher mean scores indicate greater perceived self-efficacy for screening by FIT. Change in perceived self-efficacy equals the mean at 6 months minus the mean at baseline. Change can range from -3 to 3 with positive values indicating an increase in perceived self-efficacy for screening by FIT.
Time Frame: 6 months post-baseline interview
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
Number analyzed (Participants) | 92 | 93 | 108
units on a scale | 0.07 (0.07) | 0.18 (0.07) | 0.10 (0.06)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Tailored DVD | Tailored DVD + Patient Navigation | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/123 | 4/120 | 2/128
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/120 | 0/128
Other Adverse Events (participants affected / at risk) | 0/123 | 0/120 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT03200366/Prot_SAP_000.pdf